CLINICAL TRIAL: NCT06425198
Title: A Phase 1, Multi-center, Open-label Study to Assess the Pharmacokinetics and Safety of BMS-986278 in Healthy Participants and Those With Mild, Moderate and Severe Hepatic Impairment
Brief Title: Study to Assess Drug Levels and Safety of BMS-986278 in Healthy Participants and Participants With Different Degrees of Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM027-1009
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Impairment; Healthy Participants
Keywords: Healthy Volunteers; Pharmacokinetics; Liver Diseases; Mild, Moderate and Severe Hepatic Impairment; BMS-986278
MeSH Terms: conditions — Liver Diseases; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: Mild Hepatic Impairment BMS-986278 (Experimental)
  Interventions: Drug: BMS-986278
- Group B: Moderate Hepatic Impairment BMS-986278 (Experimental)
  Interventions: Drug: BMS-986278
- Group C: Severe Hepatic Impairment BMS-986278 (Experimental)
  Interventions: Drug: BMS-986278
- Group D: Normal Hepatic Function BMS-986278 (Experimental)
  Interventions: Drug: BMS-986278

INTERVENTIONS:
Drug: BMS-986278 — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the drug levels and safety of BMS-986278 in participants with mild, moderate, and severe Hepatic Impairment (HI), and in matched healthy control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Must have a body mass index (BMI) between 18 and 40 kg/m^2 (inclusive), and body weight ≥ 50 kg.

Mild, Moderate, or Severe Hepatic Impairment Participants:

* Mild, moderate, or severe hepatic impairment (HI) or cirrhosis due to chronic hepatic disease and/or prior alcohol use.
* Mild, moderate, and severe HI participants will be enrolled according to the Child-Pugh classification score.

Matched Healthy Participants:

* Free of any clinically significant disease that would interfere with the study evaluations.
* Normal hepatic function participants will be enrolled and matched individually with HI participants with respect to age (± 10 years), weight (± 20%), sex, and race/ethnicity (Japanese and Chinese participants vs non-Japanese and non-Chinese participants).

Exclusion Criteria:

All Participants:

* History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 7 units for women, or 14 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
* Must not have had any prior exposure to BMS-986278.

Mild, Moderate, or Severe Hepatic Impairment Participants:

* Acute liver disease (eg, caused by an acute infection or drug toxicity).
* History of initial stage/planned liver transplantation within 6 months of screening or has received a liver transplant.

Matched Healthy Participants:

* Any significant medical condition, or psychiatric illness that would prevent participant from participating in the study.
* Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to day 9
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to day 9
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Up to day 9

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 62 days
Incidence of serious adverse events (SAEs) | Up to 62 days
Number of participants with physical examination abnormalities | Up to 62 days
Number of participants with vital sign abnormalities | Up to 62 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 62 days
Number of participants with clinical laboratory abnormalities | Up to 62 days
Time of maximum observed concentration (Tmax) | Up to day 9
Terminal elimination half-life (T-HALF) | Up to day 9
Apparent body clearance (CLT/F) | Up to day 9
Maximum observed plasma concentration of unbound drug (Cmax_u) | Up to day 9
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration of unbound drug [AUC(0-T)_u] | Up to day 9
Area under the plasma concentration-time curve from time 0 extrapolated to infinite time of unbound drug [AUC(INF)_u] | Up to day 9

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Local Institution - 0001, Miami Lakes, Florida
  - Local Institution - 0003, Orlando, Florida
  - Local Institution - 0002, Tampa, Florida
  - Local Institution - 0004, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com